CLINICAL TRIAL: NCT02154932
Title: Single Versus Double Dose Intra-vaginal Prostaglandin E2 "Misoprostol" Prior Abdominal Myomectomy: A Randomized Controlled Study
Brief Title: Single Versus Double Dose Intra-vaginal Prostaglandin E2 "Misoprostol" Prior Abdominal Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, ahmed M. badawy, professor, Mansoura University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AB123
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Prostaglandin E2 "Misoprostol" Prior Abdominal Myomectomy
Keywords: Myomectomy, Misoprostol
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- double dose misoprostol (Active Comparator): 2 doses, 3 and 1 hours, prior surgery (group B, 35 cases).
  Interventions: Drug: 2 doses 400 microgram misoprostol
- single dose Misoprostol (Active Comparator): intra-vaginal single dose of 400 microgram Misoprostol 1 hour pre-operatively (group A, 34 cases)
  Interventions: Drug: single dose misoprostol

INTERVENTIONS:
Drug: 2 doses 400 microgram misoprostol — 2 doses 400 microgram misoprostol, 3 and 1 hours
  Arms: double dose misoprostol
Drug: single dose misoprostol — 1 dose, 1 hours, prior surgery
  Arms: single dose Misoprostol

SUMMARY:
Introduction: The study aimed to investigate the effectiveness of a single versus double dose of Prostaglandin E2 "Misoprostol, 400 microgram" during myomectomy for multiple uterine fibroids. This was a prospective randomized controlled trial comprised of 69 patients with multiple myomas undergoing myomectomy. Patients randomly allocated to either an intra-vaginal single dose of 400 microgram Misoprostol 1 hour pre-operatively (group A, 34 cases) or 2 doses, 3 and 1 hours, prior surgery (group B, 35 cases). Operation time, intra and post-operative blood loss, hemoglobin concentration, blood pressure and body's temperature were estimated and compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients had symptomatic multiple uterine fibroids (abnormal vaginal bleeding, lower abdominal dull aching pain and pelvic heaviness, subfertility or recurrent abortion)

Exclusion Criteria:

* hypertension, cardiac and pulmonary disease, chronic endocrine or metabolic diseases such as diabetes, obesity (body mass index >30 kg/m2), all cases of single myoma and those known to be allergic to prostaglandin preparations.

Ages: 20 Years to 50 Years | Sex: Female
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
the operative time | from skin to skin in minutes
  The time from start till end of surgery
intra and post-operative blood loss | during and 6 hours after surgery
  collected soaked towels and sucked blood